CLINICAL TRIAL: NCT03078296
Title: Burnout and Associated Factors Among Members of the American Association of Gynecologic Laparoscopists
Brief Title: Burnout Among Members of AAGL
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: 111621
Record Dates: First submitted 2017-02-22; First posted 2017-03-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Members of the AAGL: Physicians and other providers who are members of the AAGL.
  Interventions: Other: survey respondents

INTERVENTIONS:
Other: survey respondents — all survey participants will be asked to complete a questionnaire

SUMMARY:
This study seeks to determine the burnout rate among minimally invasive gynecologic surgeons (MIGS) as well as to evaluate other personal, professional, and psychosocial factors associated with this condition.

An anonymous electronic survey will be sent to the American Association of Gynecologic Laparoscopists (AAGL) members. The survey will contain items that will inquire about socioeconomic background, professional characteristic, and about physical and psychologic well-being.

ELIGIBILITY:
Inclusion Criteria:

* members of the AAGL

Exclusion Criteria:

* not a member of the AAGL

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: members of the AAGL
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Burnout as assessed by questionnaire | day 1
  questionnaire assesses several factors associated with burnout including productivity and self-reported status of mental health

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States